CLINICAL TRIAL: NCT05300100
Title: Exploration of Sensory-motor Representations in Children of Typical Development Aged 5 to 8
Acronym: IMOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Lens (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-01
Record Dates: First submitted 2022-03-03; First posted 2022-03-29 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: CHILD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Activities (Experimental): The duration of the experience will last 1 hour per participant in a single session.
  The proposed actions were chosen from a very large sensorimotor repertoire of activities in everyday life for a child aged 5 to 8.
  The activities chosen involve either the whole body or specific parts such as the hand to grasp or perform graphic tests.
  Interventions: Behavioral: sensorimotor activities

INTERVENTIONS:
Behavioral: sensorimotor activities — The activities chosen involve either the whole body or specific parts such as the hand to grasp or perform graphic tests.
  * Trial 1 : Straightening: passage from sitting to sitting.
  * Trial 2 : Movement with difficulty of balance: heel-toe walking
  * Trial 3 : Movement with difficulty of balance with a structured visual environment: heel-toe walk in a contrasting fabric decoration to increase the impact of visual flow
  * Trial 4 : Move to a target, 5 m away
  * Trial 5 : Graphics: drawing of a tree. This test requires spatial skills and the establishment of median space in written transcription.
  * Trial 6 : Manual entry: collection of 12 small cubes arranged in an arc in front of the child using one hand, the choice of which will be left to the child.
  All of these tests will be offered according to a so-called "interlaced" protocol, that is to say, each execution of an action will be followed by an action simulation, and this alternation will be repeated 5 times for each task. .

SUMMARY:
Evaluate the quality of sensorimotor representations in typically developing children aged 5 to 8 years.

DETAILED DESCRIPTION:
The early coupling of perception and action makes it possible to build the sensorimotor representations, necessary for the functions of anticipation, adaptation and learning which will allow a harmonious development of motor skills throughout ontogenesis. One of the current hypotheses to explain the learning disorders detected in elementary school is a defect in the development of sensorimotor representations. Our study therefore aims to assess the quality of sensorimotor representations in typically developing children aged 5 to 8 years, using a motor imaging protocol, conventionally used in the literature in adults and patients. child. This motor imagery protocol consists of comparing the time taken by the subject to perform a given action and the time taken to imagine the action he has just performed. More precisely, the mental chronometry paradigm, based on the similarity or the difference between the two durations, makes it possible to assess the robustness of sensorimotor representations. While this isochrony is widely reported in the literature in adults, developmental studies describe onset around 9-10 years of age. Currently there is a lack of data to know the construction of these sensorimotor representations in younger children, especially during the transition to primary school. The originality of our protocol lies in two points: 1. the proposed tasks are particularly suited to young children and 2. the subject himself times his performance in the two situations: action carried out and action imagined. The duration of the experience will last 1 hour per participant in a single session.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 5 to 8
* Child enrolled in accordance with his age
* No sensory abnormality identified
* No neurodevelopmental abnormality identified

Exclusion Criteria:

* Child not affiliated to a social security scheme.
* Refusal to participate by parents and / or child

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Evaluate the quality of sensorimotor representations in typically developing children aged 5 to 8 years. | Day 1
  The primary outcome measure is the change in the gross motor imagery score. This is defined as the average of the motor imagery scores for each of the tasks performed individually;
  The motor imagery score for each individual IMtaskX task is calculated as follows:
  IMtaskX = | (DrtaskX - DitaskX) / DrtaskX |
  DrtaskX being the real measured duration of the movements performed DitaskX being the imagined duration of the movements performed Each task will be performed 5 times by each subject. DrtaskX and DitaskX are therefore an average of the 5 repetitions of the task.
  With regard to interpretation, the further the motor imagery index is from 0, the greater the difference between the duration of the imagined movement and the duration of the movement carried out, in other words the poorer the internal representations of the movement. 'action.

SECONDARY OUTCOMES:
Study the link between the construction of internal representations and overall sensorimotor skills according to age. | Day 1
  Correlation between global motor imagery score and global MABC-II score by age.
  IMtaskX = | (DrtaskX - DitaskX) / DrtaskX |
  DrtaskX being the real measured duration of the movements performed DitaskX being the imagined duration of the movements performed
Study the link between the motor imagery score of each individual task and overall sensorimotor skills by age | Day 1
  Correlation between the motor imagery score of each individual task and the overall MABC-II score by age.
  IMtaskX = | (DrtaskX - DitaskX) / DrtaskX |
  DrtaskX being the real measured duration of the movements performed DitaskX being the imagined duration of the movements performed
Study the link between the global motor imagery score, that is to say the construction of internal representations, and each of the 3 specific sensorimotor skills assessed via the MABC-II test according to age. | Day 1
  Correlation between the global motor imagery score and the individual score of each of the 3 categories of the MABC-II test according to age.
  IMtaskX = | (DrtaskX - DitaskX) / DrtaskX |
  DrtaskX being the real measured duration of the movements performed DitaskX being the imagined duration of the movements performed
Study the link between the motor imagery score of each individual task and each of the 3 sensorimotor skills assessed via the MABC-II test according to age. | Day 1
  Correlation between the motor imagery score of each individual task and the individual score of each of the 3 disciplines of the MABC-II test according to age.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Bertille DEHOUCK, Dr, Principal Investigator — Hospital of Lens
Locations (5):
- France (5):
  - Psychomotor therapist' offices, Amiens
  - Hospital Dr Schaffner, Lens
  - Hôpital Saint Vincent, Lille
  - Hospital Sambre Avesnois, Maubeuge
  - Psychomotor therapist' offices, Wavrin